CLINICAL TRIAL: NCT03610828
Title: Relation of Vegetarian Diets With Incident Cardiovascular Outcomes: A Systematic Review and Meta-analysis of Prospective Cohort Studies
Brief Title: Meta-analysis of Vegetarian Diets and Incident Cardiovascular Outcomes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, John Sievenpiper, Associate Professor, University of Toronto
Other Study IDs: DNSG-Vegetarian diets (cohort)
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Cardiovascular Diseases; Coronary Heart Disease; Stroke; Mortality
Keywords: Vegetarian Diet; Vegan Diet; Systematic Reviews and Meta-Analysis; Clinical practice guidelines; Prospective cohort studies; Cardiovascular disease; Coronary heart disease; Stroke; Cardiovascular mortality; Coronary heart disease mortality; Stroke mortality
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Stroke | interventions — Diet, Vegan

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Vegetarian or Vegan Diets — Diets that omit all animal products (vegan diet) or all animal products with the exception of eggs and/or dairy products (vegetarian)

SUMMARY:
Vegetarian and vegan diets have been shown to reduce cardiometabolic risk factors for chronic diseases, such as cardiovascular disease and diabetes, and have been associated with decreased risk of these chronic diseases. The role of vegetarian and/or vegan dietary patterns and incident cardiovascular outcomes still remains unclear. To address these uncertainties, the investigators propose to conduct a systematic review and meta-analysis of the totality of evidence from prospective cohort studies to distinguish the association of vegetarian and/or vegan dietary patterns on the prevention and management of cardiovascular diseases. This proposed knowledge synthesis was commissioned by the Diabetes and Nutrition Study Group (DNSG) of the European Association for the Study of Diabetes (EASD) and will be used to inform clinical practice and dietary guidelines, help improve health outcomes, and guide future research design.

DETAILED DESCRIPTION:
Background: Cardiovascular disease (CVD) is the number 1 cause of death worldwide, representing 31% of all deaths. Vegetarian and/or vegan dietary patterns have been shown in prospective cohort and cross-sectional studies to be associated with lower coronary heart disease and ischemic heart disease risk. Evidence from randomized controlled trials also suggest that vegetarian and vegan diets may be beneficial for cardiovascular disease risk factors, such as LDL cholesterol, weight, blood pressure and type 2 diabetes (glycemic control). Moreover, evidence from meta-analyses of prospective cohort studies have shown that diets high in red and processed meat consumption are associated with an increased incidence of stroke and cardiovascular mortality. The evidence for a vegetarian dietary pattern is promising for prevention and management of cardiovascular diseases, however, not all CVD guidelines recommend following a vegetarian and/or vegan dietary pattern for the prevention and management of these diseases, or the guidelines grade the evidence as low quality.

Need for proposed research: High quality systematic reviews and meta-analyses of prospective cohort studies represent evidence to support dietary guidelines and public health policy development. As dietary guidelines and public health policy have shifted toward food and dietary-pattern based recommendations, there is a need for systematic reviews and meta-analyses comparing the role of vegetarian/vegan diets in the prevention and management of cardiovascular diseases.

Objective: The investigators will conduct a systematic reviews and meta-analysis to assess vegan/vegetarian diets with cardiovascular disease outcomes (cardiovascular disease (CVD), coronary heart disease (CHD) and stroke incidence and mortality) in prospective cohort studies.

Design: The planning and conduct of the proposed meta-analyses will follow the Cochrane handbook for systematic reviews of interventions. The reporting will follow the Meta-analysis Of Observational Studies in Epidemiology (MOOSE) guidelines.

Data sources: MEDLINE, EMBASE, and The Cochrane Central Register of Controlled Trials databases will be searched using appropriate search terms supplemented by hand searches of references of included studies.

Data extraction: Two or more investigators will independently extract relevant data and assess risk of bias using the Newcastle-Ottawa Scale (NOS) for observational studies. Risk ratios, odds ratios and hazard ratios for clinical outcomes will be extracted or derived from clinical event data across exposure to either vegetarian or non-vegetarian diets. All disagreements will be resolved by consensus.

Outcomes: Six outcomes will be assessed: CVD incidence and mortality, coronary heart disease (CHD) incidence and mortality, stroke incidence and mortality

Data synthesis: The natural log-transformed relative risks or hazard ratios of clinical outcomes comparing the exposure to the reference group from each cohort will be pooled using the generic inverse variance method with random effects models. Heterogeneity will be assessed by Cochrane's Q and quantified by I2. Sensitivity analyses and a priori subgroup analyses will be undertaken to explore sources of heterogeneity including the effect of the cohorts, sex, type of vegetarian diet, underlying disease status, follow-up (<10-years, >=10-years), level of adjustment of models, quality of the studies (NOS), and validation of the dietary assessment instruments. Significant unexplained heterogeneity will be investigated by additional post hoc subgroup analyses. Meta-regression analyses will assess the significance of subgroups analyses. Publication bias will be assessed by the inspection of funnel plots and using Begg's and Egger's tests.

Evidence Assessment: The certainty of the evidence for each outcome will be assessed using the Grading of Recommendations Assessment, Development and Evaluation (GRADE).

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition, cardiovascular diseases and diabetes. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined. Applicant/Co-applicant Decision Makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

Significance: The proposed project will aid in knowledge translation related to the role of vegetarian/vegan diets in the prevention and management of cardiovascular diseases, strengthening the evidence-base for guidelines and improving health outcomes by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

ELIGIBILITY:
Inclusion Criteria:

* Prospective cohorts studies
* Duration >=1 year
* Assessment of the exposure of vegetarian or vegan diet
* Ascertainment of viable data by level of exposure

Exclusion Criteria:

* Ecological, cross-sectional, retrospective observational studies, clinical trials and non-human studies
* Duration < 1 year
* No assessment of exposure of vegetarian/vegan diet
* No ascertainment viable clinical outcome data by level of exposure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers or those at risk for cardiovascular disease
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular disease incidence | Up to 20 years
Cardiovascular disease mortality | Up to 20 years
Coronary heart disease incidence | Up to 20 years
Coronary heart disease mortality | Up to 20 years
Stroke incidence | Up to 20 years
Stroke mortality | Up to 20 years

CONTACTS AND LOCATIONS:
Overall Officials: John Sievenpiper, PhD, MD, Principal Investigator — University of Toronto
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Satija A, Bhupathiraju SN, Spiegelman D, Chiuve SE, Manson JE, Willett W, Rexrode KM, Rimm EB, Hu FB. Healthful and Unhealthful Plant-Based Diets and the Risk of Coronary Heart Disease in U.S. Adults. J Am Coll Cardiol. 2017 Jul 25;70(4):411-422. doi: 10.1016/j.jacc.2017.05.047. PMID 28728684
- [Background] World Health Organization. (2017). Cardiovascular Diseases. Obtained from: http://www.who.int/mediacentre/factsheets/fs317/en/
- [Background] Dinu M, Abbate R, Gensini GF, Casini A, Sofi F. Vegetarian, vegan diets and multiple health outcomes: A systematic review with meta-analysis of observational studies. Crit Rev Food Sci Nutr. 2017 Nov 22;57(17):3640-3649. doi: 10.1080/10408398.2016.1138447. PMID 26853923
- [Background] Barnard ND, Cohen J, Jenkins DJ, Turner-McGrievy G, Gloede L, Jaster B, Seidl K, Green AA, Talpers S. A low-fat vegan diet improves glycemic control and cardiovascular risk factors in a randomized clinical trial in individuals with type 2 diabetes. Diabetes Care. 2006 Aug;29(8):1777-83. doi: 10.2337/dc06-0606. PMID 16873779
- [Background] Barnard ND, Cohen J, Jenkins DJ, Turner-McGrievy G, Gloede L, Green A, Ferdowsian H. A low-fat vegan diet and a conventional diabetes diet in the treatment of type 2 diabetes: a randomized, controlled, 74-wk clinical trial. Am J Clin Nutr. 2009 May;89(5):1588S-1596S. doi: 10.3945/ajcn.2009.26736H. Epub 2009 Apr 1. PMID 19339401
- [Background] Mishra S, Xu J, Agarwal U, Gonzales J, Levin S, Barnard ND. A multicenter randomized controlled trial of a plant-based nutrition program to reduce body weight and cardiovascular risk in the corporate setting: the GEICO study. Eur J Clin Nutr. 2013 Jul;67(7):718-24. doi: 10.1038/ejcn.2013.92. Epub 2013 May 22. PMID 23695207
- [Background] Wang X, Lin X, Ouyang YY, Liu J, Zhao G, Pan A, Hu FB. Red and processed meat consumption and mortality: dose-response meta-analysis of prospective cohort studies. Public Health Nutr. 2016 Apr;19(5):893-905. doi: 10.1017/S1368980015002062. Epub 2015 Jul 6. PMID 26143683
- [Background] Yang C, Pan L, Sun C, Xi Y, Wang L, Li D. Red Meat Consumption and the Risk of Stroke: A Dose-Response Meta-analysis of Prospective Cohort Studies. J Stroke Cerebrovasc Dis. 2016 May;25(5):1177-1186. doi: 10.1016/j.jstrokecerebrovasdis.2016.01.040. Epub 2016 Feb 27. PMID 26935118
- [Background] Coutts SB, Wein TH, Lindsay MP, Buck B, Cote R, Ellis P, Foley N, Hill MD, Jaspers S, Jin AY, Kwiatkowski B, MacPhail C, McNamara-Morse D, McMurtry MS, Mysak T, Pipe A, Silver K, Smith EE, Gubitz G; Heart, and Stroke Foundation Canada Canadian Stroke Best Practices Advisory Committee. Canadian Stroke Best Practice Recommendations: secondary prevention of stroke guidelines, update 2014. Int J Stroke. 2015 Apr;10(3):282-91. doi: 10.1111/ijs.12439. Epub 2014 Dec 23. PMID 25535808
- [Background] Anderson TJ, Gregoire J, Pearson GJ, Barry AR, Couture P, Dawes M, Francis GA, Genest J Jr, Grover S, Gupta M, Hegele RA, Lau DC, Leiter LA, Lonn E, Mancini GB, McPherson R, Ngui D, Poirier P, Sievenpiper JL, Stone JA, Thanassoulis G, Ward R. 2016 Canadian Cardiovascular Society Guidelines for the Management of Dyslipidemia for the Prevention of Cardiovascular Disease in the Adult. Can J Cardiol. 2016 Nov;32(11):1263-1282. doi: 10.1016/j.cjca.2016.07.510. Epub 2016 Jul 25. PMID 27712954
- [Derived] Glenn AJ, Viguiliouk E, Seider M, Boucher BA, Khan TA, Blanco Mejia S, Jenkins DJA, Kahleova H, Rahelic D, Salas-Salvado J, Kendall CWC, Sievenpiper JL. Relation of Vegetarian Dietary Patterns With Major Cardiovascular Outcomes: A Systematic Review and Meta-Analysis of Prospective Cohort Studies. Front Nutr. 2019 Jun 13;6:80. doi: 10.3389/fnut.2019.00080. eCollection 2019. PMID 31263700